CLINICAL TRIAL: NCT05798702
Title: Fibrosis Reduction in Non Alcoholic Steatohepatitis: the Effects of Weight Loss vs Metabolic Surgery
Brief Title: Fibrosis Reduction in Non Alcoholic Steatohepatitis
Acronym: FRIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mingrone Geltrude, professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4103
Record Dates: First submitted 2023-02-16; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: NASH With Fibrosis; Weight Loss; Bariatric Surgery Candidate
MeSH Terms: conditions — Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive lifestyle modifications (Active Comparator): VLCD 800-850 Kcal/day
  Interventions: Dietary Supplement: intensive life style modification
- Roux-en-y-gastric bypass (Active Comparator): laparoscopic RYGB
  Interventions: Procedure: roux -en-y- gastric bypass

INTERVENTIONS:
Procedure: roux -en-y- gastric bypass — Roux-&-Y Gastric Bypass (RYGB) involves the use of a surgical stapler to create a small and vertically oriented gastric pouch with a volume of 30 ml. The upper pouch is completely divided by the gastric remnant and is anastomosed to the jejunum, 75 cm distally to the Treitz's ligament, through a narrow gastrojejunal anastomosis in a Roux-en-Y fashion. Bowel continuity is restored by an entero-entero anastomosis, between the excluded biliary limb and the alimentary limb, performed at 100 cm from the gastrojejunostomy.
  Arms: Roux-en-y-gastric bypass
Dietary Supplement: intensive life style modification — Weight loss will be induced using a VLCD (800-850 kcal/day; 59% carbohydrate, 13% fat, 26% protein, 2% fiber) with replacement meals for 2 months, followed by structured food reintroduction every 2-8 weeks (about 50% carbohydrate, 35% total fat, and 15% protein), and an ongoing structured program with follow-up visits up to 25% body weight loss
  Arms: intensive lifestyle modifications

SUMMARY:
Background: Non-Alcoholic Steatohepatitis (NASH) represents one of the stages of Non-Alcoholic Fatty Liver Disease (NAFLD) with a very high risk to evolve in cirrhosis and hepato-carcinoma.

Currently, the only diagnostic method is a liver biopsy that remains the gold standard for characterizing liver histologic alterations and fibrosis stages. There is no specific treatment for NASH, in fact no drugs are currently licensed specifically for treating this disease.

Aim: Our aim is to conduct a non-inferiority, randomized-controlled trial (RCT) comparing Roux-en-Y Gastric bypass (RYGB) with an intensive lifestyle modification plan (Very low-calorie diet, VLCD) for the reduction of advanced stages of fibrosis in subjects with obesity and NASH after 25% weight loss.

DETAILED DESCRIPTION:
Materials and Methods: The Investigators will screen patients with obesity, NAFLD fibrosis score (NFS) >0.676 and FibroScan > 9.5 kPA who have a high probability of NASH with advanced stage of fibrosis.

Participants will undergo liver biopsy to make diagnosis according to the Steatosis Activity Fibrosis (SAF) score algorithm. Subjects with BMI ≥ 30 and ≤50 kg/m2, age 25-65 years and F3-F4 fibrosis stage at liver biopsy will be included and randomized 1:1 to RYGB or VLCD. Anthropometric parameters, body composition with DEXA and liver function with blood samples will be assessed at the enrolment. A mixed meal metabolic test will be also performed to evaluate insulin sensitivity and secretion. These procedures will be repeated after 25% weight loss. Expectation: The Investigators expect a reduction of 2 points of histological fibrosis after 25% weight loss following either metabolic surgery or dieting. The investigators foresee also reversal of NASH, improvement of metabolic syndrome and glycemic control, changes in insulin sensitivity and secretion, changes in lipid profile, in NASH liver markers, in Fibroscan variables and in body composition

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed before starting any procedure foreseen by the study;
* Liver Ultrasound shoving steatosis and Fibroscan>9,5 KPa;
* NAFLD fibrosis score>0,676;
* diagnosis of NASH with stage F3-F4 of fibrosis according to SAF score, documented by liver biopsy and no evidence of another form of liver disease;
* BMI≥ 30 and ≤50 kg/m2;
* Age 25-65 years.

Exclusion Criteria:

* Chronic liver disease other than NAFLD (e.g. hemochromatosis, viral or autoimmune hepatitis, Wilson's disease, α1 -antitrypsin deficiency);
* Presence of esophageal varices and/or ascites;
* INR ≥ 1,4;
* Platelet count ≤ 100000;
* Substantial alcohol consumption (>20 g/day for women or >30 g/day for men) and/or toxin exposure;
* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous 6 months;
* End stage renal failure;
* Participation in any other concurrent therapeutic clinical trial;
* Any other life-threatening, non-cardiac disease;
* Pregnancy;
* Type 1 diabetes, or LADA;
* Lipodystrophy;
* Abetalipoproteinemia;
* Interfering medications (e.g., amiodarone, methotrexate, tamoxifen, corticosteroids);
* Inability to give informed consent.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
histological reduction of fibrosis | 2 years
  The primary outcome is the rate of histological reduction of 2 points of fibrosis after 25% weight loss following either metabolic surgery or dieting

SECONDARY OUTCOMES:
Liver histology | 2 years
  Reversal of NASH: number of partcipant with a NAFLD activity score (NAS: from 0 to 8) < 3;
  Changes in Fibroscan evaluation: number of participant with a FibroScan <9.5 kPa.
Liver Markers | 2 years
  Changes in liver markers: number of participant with a significant reduction of AST and ALT from baseline;
Non-alcoholic Fatty Liver Disease Fibrosis score | 2 years
  Changes in Non-alcoholic Fatty Liver Disease Fibrosis score from baseline
Fibrosis-4 (FIB-4) Index | 2 years
  Changes in Fibrosis-4 (FIB-4) Index for Liver Fibrosis from baseline;
Fibroscan | 2 years
  Changes in Fibroscan evaluation: number of participant with a FibroScan <9.5 kPa.

CONTACTS AND LOCATIONS:
Overall Officials: geltrude mingrone, professor, Principal Investigator — Policlinico A. Gemelli IRCCS
Locations (1):
- Mingrone Geltrude, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Younossi ZM. Non-alcoholic fatty liver disease - A global public health perspective. J Hepatol. 2019 Mar;70(3):531-544. doi: 10.1016/j.jhep.2018.10.033. Epub 2018 Nov 9. PMID 30414863
- [Result] Vilar Gomez E, Rodriguez De Miranda A, Gra Oramas B, Arus Soler E, Llanio Navarro R, Calzadilla Bertot L, Yasells Garcia A, Del Rosario Abreu Vazquez M. Clinical trial: a nutritional supplement Viusid, in combination with diet and exercise, in patients with nonalcoholic fatty liver disease. Aliment Pharmacol Ther. 2009 Nov 15;30(10):999-1009. doi: 10.1111/j.1365-2036.2009.04122.x. Epub 2009 Aug 18. PMID 19691668
- [Result] Dixon JB, Bhathal PS, Hughes NR, O'Brien PE. Nonalcoholic fatty liver disease: Improvement in liver histological analysis with weight loss. Hepatology. 2004 Jun;39(6):1647-54. doi: 10.1002/hep.20251. PMID 15185306
- [Result] Glass LM, Dickson RC, Anderson JC, Suriawinata AA, Putra J, Berk BS, Toor A. Total body weight loss of >/= 10 % is associated with improved hepatic fibrosis in patients with nonalcoholic steatohepatitis. Dig Dis Sci. 2015 Apr;60(4):1024-30. doi: 10.1007/s10620-014-3380-3. Epub 2014 Oct 30. PMID 25354830
- [Result] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Nanni G, Castagneto M, Bornstein S, Rubino F. Bariatric-metabolic surgery versus conventional medical treatment in obese patients with type 2 diabetes: 5 year follow-up of an open-label, single-centre, randomised controlled trial. Lancet. 2015 Sep 5;386(9997):964-73. doi: 10.1016/S0140-6736(15)00075-6. PMID 26369473
- [Result] Lassailly G, Caiazzo R, Buob D, Pigeyre M, Verkindt H, Labreuche J, Raverdy V, Leteurtre E, Dharancy S, Louvet A, Romon M, Duhamel A, Pattou F, Mathurin P. Bariatric Surgery Reduces Features of Nonalcoholic Steatohepatitis in Morbidly Obese Patients. Gastroenterology. 2015 Aug;149(2):379-88; quiz e15-6. doi: 10.1053/j.gastro.2015.04.014. Epub 2015 Apr 25. PMID 25917783
- [Result] Lassailly G, Caiazzo R, Ntandja-Wandji LC, Gnemmi V, Baud G, Verkindt H, Ningarhari M, Louvet A, Leteurtre E, Raverdy V, Dharancy S, Pattou F, Mathurin P. Bariatric Surgery Provides Long-term Resolution of Nonalcoholic Steatohepatitis and Regression of Fibrosis. Gastroenterology. 2020 Oct;159(4):1290-1301.e5. doi: 10.1053/j.gastro.2020.06.006. Epub 2020 Jun 15. PMID 32553765
- [Result] Vilar-Gomez E, Martinez-Perez Y, Calzadilla-Bertot L, Torres-Gonzalez A, Gra-Oramas B, Gonzalez-Fabian L, Friedman SL, Diago M, Romero-Gomez M. Weight Loss Through Lifestyle Modification Significantly Reduces Features of Nonalcoholic Steatohepatitis. Gastroenterology. 2015 Aug;149(2):367-78.e5; quiz e14-5. doi: 10.1053/j.gastro.2015.04.005. Epub 2015 Apr 10. PMID 25865049
- [Result] Bedossa P, Poitou C, Veyrie N, Bouillot JL, Basdevant A, Paradis V, Tordjman J, Clement K. Histopathological algorithm and scoring system for evaluation of liver lesions in morbidly obese patients. Hepatology. 2012 Nov;56(5):1751-9. doi: 10.1002/hep.25889. PMID 22707395
- [Result] Angulo P, Hui JM, Marchesini G, Bugianesi E, George J, Farrell GC, Enders F, Saksena S, Burt AD, Bida JP, Lindor K, Sanderson SO, Lenzi M, Adams LA, Kench J, Therneau TM, Day CP. The NAFLD fibrosis score: a noninvasive system that identifies liver fibrosis in patients with NAFLD. Hepatology. 2007 Apr;45(4):846-54. doi: 10.1002/hep.21496. PMID 17393509
- [Result] de Almeida SR, Rocha PR, Sanches MD, Leite VH, da Silva RA, Diniz MT, Diniz Mde F, Rocha AL. Roux-en-Y gastric bypass improves the nonalcoholic steatohepatitis (NASH) of morbid obesity. Obes Surg. 2006 Mar;16(3):270-8. doi: 10.1381/096089206776116462. PMID 16545157